CLINICAL TRIAL: NCT03178916
Title: Breast Feeding Practice in High Risk Pregnant Women
Status: Completed | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Ahmed Mohamed Abbas, principal investigator, Assiut University
Other Study IDs: BFHRP
Record Dates: First submitted 2017-06-06; First posted 2017-06-07 (Actual); Last update posted 2021-04-23 (Actual); Status verified 2021-04

CONDITIONS: Breast Feeding
MeSH Terms: conditions — Breast Feeding

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Low risk pregnant women: evaluation of the efficacy of breastfeeding Low risk pregnant women
- high risk pregnant women: evaluation of the efficacy of breastfeeding high risk pregnant women

SUMMARY:
The American Academy of Paediatrics recognizes multiple benefits of breastfeeding to both the term and premature newborn, particularly with regard to protection from infectious agents. Studies have demonstrated decreased rates of bacteraemia, meningitis, respiratory and urinary tract infections, necrotizing enterocolitis, and otitis media among breastfed infants

ELIGIBILITY:
Inclusion Criteria:

1. Diabetes mellitus.
2. Cardiac disease.
3. Essential hypertension.
4. Chronic chest disease, and/or chronic TB infection.
5. Chronic hepatitis.
6. Neurologic disease.
7. Anaemia (Hemoglobin <10 gm/dL).
8. Thyroid disease.
9. Multiple pregnancy.

Exclusion Criteria:

* pregnant women < 34 weeks.

Ages: 20 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: Patients attending Sohag general hospital
Sampling Method: Probability Sample
Enrollment: 140 (Actual)
Dates: Start 2017-07-01 (Actual); Primary Completion 2020-10-31 (Actual); Study Completion 2020-12-31 (Actual)

PRIMARY OUTCOMES:
The number of breast feeding women during pregnancy | 6 months

CONTACTS AND LOCATIONS:
Locations (1):
- Assiut Faculty of Medicine, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: No